CLINICAL TRIAL: NCT06455787
Title: J-Valve to Treat Aortic Regurgitation Via Transcatheter Therapy
Brief Title: J-Valve Transfemoral Pivotal Study
Acronym: JOURNEY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JC Medical, Inc., an affiliate of Edwards Lifesciences LLC (Industry)
Collaborators: Minneapolis Heart Institute Foundation (Other); Cardiovascular Research Foundation, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JCM-002
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-08

CONDITIONS: Aortic Valve Regurgitation; Aortic Valve Disease Mixed
Keywords: J-Valve Transfemoral System; Transcatheter Therapy; Transcatheter Aortic Valve Replacement; TAVR; Transfemoral
MeSH Terms: conditions — Aortic Valve Insufficiency | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: The investigation is a prospective, single arm, multi-center, interventional pivotal study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- J-Valve Transfemoral (TF) System (Experimental)
  Interventions: Device: J-Valve Transfemoral (TF) System

INTERVENTIONS:
Device: J-Valve Transfemoral (TF) System — Treatment includes using the J-Valve Transfemoral (TF) System, a transcatheter aortic valve replacement system that consists of the J-Valve TF Bioprosthesis and the J-Valve TF Delivery Device and Loading Accessories, during transcatheter aortic valve replacement (TAVR). The Edwards 16Fr eSheath+ Introducer Set may be used for the introduction and removal of the J-Valve TF System.

SUMMARY:
The primary objective of this study is to assess the safety and efficacy of the J-Valve Transfemoral (TF) System in patients with symptomatic, severe (grade 3 or 4), native aortic valve regurgitation (AR) and AR-dominant mixed aortic valve disease, who are judged by a multi-disciplinary heart team to be at high risk for open surgical aortic valve replacement (SAVR).

A Cardiac Magnetic Resonance (CMR) sub-study will examine if intervention for AR translates to improved ventricular remodeling, the impact of LV remodeling on clinical outcomes and quality of life, as well as volumetric and myocardial differences between genders.

DETAILED DESCRIPTION:
This is a prospective, single arm, multi-center, interventional pivotal study that will enroll up to 194 subjects in up to 35 investigational sites, predominantly in the United States and up to 7 in Canada, Europe, and Japan. Of the 194 subjects, the CMR imaging sub-study will include up to 75 subjects with severe AR already confirmed by TTE. Additionally, up to 40 roll-in subjects may be treated to enable clinical experience and exposure to the device while allowing a reasonable learning curve. The subjects will then be followed 5-years post-procedure of the J-Valve TF System.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic according to New York Heart Association (NYHA) functional class (FC) II or higher
2. Severe AR, defined as follows, as assessed by Imaging Core Laboratory:

   A. Severe AR by Transthoracic Echocardiography (TTE) (grade 3 or 4)

   B. OR, if indeterminate AR, by TTE, ANY ONE of the following:

   i. Cardiac magnetic resonance imaging (CMR)-derived aortic regurgitant fraction (RF) ≥43% ii. CMR-derived RF ≥33% + left ventricular dilation (left ventricular end diastolic volume index [LVEDVi]) >105 mL/m^2 for men or LVEDVi >96 mL/m^2 for women) iii. CMR-derived RF ≥33% + LV ejection fraction (LVEF) ≤55% or left ventricular end systolic volume index (LVESVi) ≥43mL/m^2; iv. Severe AR by Transesophageal Echocardiography (TEE) (grade 3 or 4)
3. High risk for surgery as judged by a multi-disciplinary heart team
4. Suitable anatomy to accommodate the insertion, delivery, and deployment of the study devices (see anatomic exclusions below)
5. Written informed consent and agreement to comply with all required post-procedure follow-up visits at investigational site.

Exclusion Criteria:

1. Previous prosthetic aortic valve (bioprosthesis or mechanical) implant
2. Aortic valve stenosis > moderate*
3. Severe mitral valve or tricuspid valve regurgitation*
4. Severe mitral valve or tricuspid valve stenosis*
5. Active infection, including infective endocarditis
6. Cardiac imaging evidence of cardiac mass, thrombus or vegetation
7. Inability to tolerate or a condition precluding treatment with antithrombotic (antiplatelet, anticoagulant) therapy
8. Renal insufficiency (eGFR <30 mL/min/1.73m^2) or end stage renal disease requiring chronic dialysis
9. Liver disease (cirrhosis of the liver [Child-Pugh Class B or C])
10. Blood dyscrasias as defined: leukopenia (WBC <3000 cells/mcL), thrombocytopenia (platelet count <50,000 cells/mcL), anemia (hemoglobin <9 g/dL), history of bleeding diathesis coagulopathy, or hypercoagulable state (unless therapeutically stable)
11. Known hypersensitivity or contraindication to aspirin, heparin, bivalirudin, clopidogrel, Nitinol (Nickel, Titanium) or sensitivity to contrast media, which cannot be adequately premedicated
12. Left ventricular dysfunction with left ventricular ejection fraction (LVEF) <25% as measured by resting echocardiogram (or by CMR, when performed)*
13. Clinically significant untreated coronary artery disease requiring revascularization or anticipated coronary revascularization procedure within 12-months post index procedure
14. Acute myocardial infarction within 30 days prior to index procedure
15. PCI within 30 days prior to index procedure
16. Carotid intervention within 6 weeks prior to index procedure or carotid artery disease requiring intervention
17. Previous, or planned, other surgical or interventional procedures within 30 days before, during, or within 30 days after the index procedure
18. Uncontrolled atrial fibrillation
19. Severe right ventricular (RV) dysfunction*
20. Pulmonary hypertension (systolic PA pressure >70mmHg or systolic PA pressure ≥2/3 of systemic systolic BP)
21. Severe chronic obstructive pulmonary disease (COPD) requiring chronic oral steroids or requiring continuous home O2
22. Stroke (CVA), transient ischemic attack (TIA) or neurological signs and symptoms attributed to carotid or vertebrobasilar disease within 90 days prior to index procedure
23. Cardiogenic shock defined as systolic blood pressure <90 mmHg in addition to signs of tissue hypoperfusion or the need for vasopressors and/or mechanical hemodynamic support to maintain systolic blood pressure ≥90mmHg
24. Patient requires mechanical circulatory support within 30 days prior to index procedure
25. Estimated life expectancy of less than 24 months due to associated non-cardiac co-morbid conditions
26. Pregnancy or intent to become pregnant prior to completion of all protocol follow-up requirements
27. Participation in another investigational study that has not reached its primary endpoint
28. Considered to be part of a vulnerable population

    * As assessed by Imaging Core Laboratory

Anatomic Exclusions:

1. Ascending Aortic diameter >5 cm*
2. Aortic Annulus Perimeter <57 mm or >104 mm*
3. Inappropriate anatomy for femoral introduction and delivery of the study system
4. Left ventricular end-diastolic diameter (LVEDD) >75 mm*
5. Congenital aortic valve disease including Unicuspid, Bicuspid, or Quadricuspid aortic valve anatomy*
6. Congenital univentricle or other condition that, in the opinion of the investigator and/or consulting physician, may constitute an unwarranted surgical risk
7. Excessive aortic valve prolapse that would preclude proper seating of the implant in the aortic annulus
8. Abdominal/thoracic aortic aneurysm ≥5.0 cm*
9. Aorto-iliac disease requiring intervention to facilitate delivery of access sheath
10. Excessive tortuosity of delivery system pathway, defined as severe tortuosity of multiple vessels including iliofemoral, thoracoabdominal aorta, aortic arch, or LV-aortic root angle >80⁰

    * As assessed by Imaging Core Laboratory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at 1 year | 1-year post-procedure
The composite rate of early-safety outcomes at 30 days as defined by the Valve Academic Research Consortium 3 (VARC-3) | 30-days post-procedure
  Includes:
  * All-cause death
  * All stroke
  * VARC-3 type 2-4 bleeding
  * Major vascular, access-related, or cardiac structural complication
  * Acute kidney injury (AKI) stage 3 or 4
  * New permanent pacemaker due to procedure-related conduction abnormalities
  * Surgery or intervention related to the device

SECONDARY OUTCOMES:
Rate of improvement in cardiovascular-specific health status | Baseline to 1-year follow-up
  As measured by the Kansas City Cardiomyopathy Questionnaire overall summary score (KCCQ-OS)
Improvement in left ventricular end diastolic diameter index (LVEDDi) | Baseline to 1-year follow-up
  To measure LV remodeling
Improvement in left ventricular end diastolic volume index (LVEDVi) | Baseline to 1-year follow-up
  To measure LV remodeling
Improvement in effective stroke volume index (ESVi) | Baseline to 1-year follow-up
  To measure LV remodeling
Improvement in effective cardiac output index (ECOi) | Baseline to 1-year follow-up
  To measure LV remodeling

CONTACTS AND LOCATIONS:
Overall Officials: Dean J Kereiakes, MD, Study Chair — The Christ Hospital Heart & Vascular Institute; Michael Reardon, MD, Study Chair — The Methodist Hospital Research Institute; Santiago Garcia, MD, Principal Investigator — The Christ Hospital and The Carl and Edyth Lindner Center for Research and Education; Tsuyoshi Kaneko, MD, Principal Investigator — Washington University School of Medicine
Locations (31):
- United States (31):
  - HonorHealth Research & Innovation Institute, Scottsdale, Arizona
  - Cedars Sinai, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Bay Area Structural Heart at Sutter Health, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - UC Health Northern Colorado (Medical Center of the Rockies), Loveland, Colorado
  - NCH Rooney Heart Institute, Naples, Florida
  - Emory University Atlanta, Atlanta, Georgia
  - Piedmont, Atlanta, Georgia
  - Northwestern University Chicago, Chicago, Illinois
  - Glenbrook - Endeavor Health, Glenview, Illinois
  - Ascension Via Christi, Wichita, Kansas
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Massachusetts General Hospital Boston, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital Detroit, Detroit, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - CentraCare Heart and Vascular Center, Saint Cloud, Minnesota
  - Washington University - Barnes-Jewish Hospital St. Louis, St Louis, Missouri
  - University at Buffalo - Kaleida Health, Buffalo, New York
  - Columbia University Irving Medical Center/New York-Presbyterian Hospital, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - The Lindner Research Center at The Christ Hospital, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Ascension St. Thomas West Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - HCA Houston Healthcare Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - The Heart Hospital - Baylor Plano, Plano, Texas
  - Swedish Heart & Vascular Research, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No